CLINICAL TRIAL: NCT06272305
Title: TREC - Evaluation of the Impact of Eversion Technical Features on the Rate of Carotid Restenosis
Acronym: TREC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Principal Investigator, Nicolas RIFFET-VIDAL, Research and Innovation Director, University Hospital, Angers
Other Study IDs: 49RC21_0301
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Hyperplasia
MeSH Terms: conditions — Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: This research does not require any specific investigation and does not imply any modification of treatment. — Collection of data from the medical record for patients with a non specific carotid endarterectomy

SUMMARY:
Restenosis due to myo-intimal hyperplasia remains a concern after carotid endarterectomy. It occurs in around 6% of cases. Several risk factors for restenosis have already been identified, such as smoking, hypertension, female gender, diabetes, dyslipidemia and small carotid diameter. The main objective of this prospective multicenter study was to determine whether the technical characteristics of the eversion technique have an influence on the rate of restenosis at 1 year.

Between September 2021 and November 2022, we followed all patients undergoing carotid endarterectomy by eversion in 8 French hospitals. Demographic data, operative indications and technical characteristics of the endarterectomies performed were collected. These were defined by the circumferential nature of the carotid bulb according to 3 types (TREC A, B or C), and the length and depth of the endarterectomy according to anatomopathological reports. Post-operative complications were collected as much as doppler ultrasonography at three months and 1 year to quantify restenosis.

DETAILED DESCRIPTION:
Before the surgery, the following data is collected :

* General data: Sex, age, weight, height
* History and cardiovascular risk factors: diabetes, high blood pressure, dyslipidemia, smoking, chronic renal failure, etc.
* Current treatments taken by the patient
* The degree of initial stenosis of the carotid artery of interest on duplex ultrasound as well as on CT angiography
* The context of endarterectomy if it occurs following a stroke or preventively.

Data to be recovered post-operatively from carotid surgery :

* The operative report specifying the circumferential nature of the carotid endarterectomy on the common carotid-external carotid axis.

  3 possible categories: no endarterectomy, non-circumferential partial endarterectomy, circumferential endarterectomy.
* Post-operative doppler (< 1 month) assessing the presence of residual stenosis.
* The patient's operative consequences with the occurrence of intercurrent cardiological events (cardiological, biological or electrocardiographic), neurological (central or peripheral), post-operative complications such as cervical hematoma.

Visit between month 1 and month 3 :

* The anatomopathological report specifying: Length of the endarterectomy part in millimeters and the depth of the endarterectomy according to the location of the separation plane at the level of the artery wall (deep or superficial intimal plane).
* Doppler assessing the presence of carotid restenosis
* The occurrence of central neurological events that may be related to the endarterectomized carotid artery

Visit at one year :

* Doppler assessing the presence of carotid restenosis
* The occurrence of central neurological events that may be related to the endarterectomized carotid artery

ELIGIBILITY:
Inclusion Criteria:

Any patient who is having carotid endarterectomy by eversion according to HAS + ESVS recommendations :

* Stenosis > 70% on dopplerin the absence of neurological symptoms attributable to the carotid territory affected by the stenotic artery.
* Stenosis > 50% with neurological symptoms attributable to the carotid territory affected by the stenotic artery.

Exclusion Criteria:

* Any carotid revascularization technique other than eversion (carotid endarterectomy with patch, carotid resection-anastomosis or bypass).
* Cardiac surgery combined with carotid surgery
* Minor patients
* Endovascular carotid surgery
* Opposition to use patient's data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who is having carotid endarterectomy by eversion
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of restenosis | one year
  The main objective is to evaluate the rate of restenosis at doppler(defined as restenosis ≥50%(NASCET/ECST)) occurring at one year, according to the technical characteristics of the eversion. They are defined according to three distinct criteria: the circumferential nature of the endarterectomy at the level of the carotid bifurcation, the length of the endarterectomy and its depth in the plane of the intima.

SECONDARY OUTCOMES:
Morbidity and mortality rate | 30 days
  Cumulative morbidity and mortality rate at 30 days defined by:
  * All-cause mortality within 30 days post-op
  * Major neurological event defined as the occurrence of a stroke (focal signs lasting more than 24 hours, confirmed by brain imaging)
Major cardiological event | one year
  Major cardiological event defined by troponin elevation with chest pain (or equivalent symptom) and/or ECG changes in favor of myocardial ischemia
Minor neurological events | one year
  Minor neurological events: peripheral neurological and/or cranial nerve damage (tongue deviation, dysphonia, swallowing disorder).

CONTACTS AND LOCATIONS:
Overall Officials: Gautier HAUPERT, Dr, Principal Investigator — university hospital of Angers

IPD SHARING:
Plan to Share IPD: No